CLINICAL TRIAL: NCT04816916
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of AXA1665 in Subjects With Liver Cirrhosis and Prior Overt Hepatic Encephalopathy (EMMPOWER)
Brief Title: Efficacy and Safety of AXA1665 in Cirrhotic Subjects With Prior Overt Hepatic Encephalopathy
Acronym: EMMPOWER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor is stopping the study to focus company resources on other development programs.
Sponsor: Axcella Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXA1665-101
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Hepatic Encephalopathy
Keywords: liver cirrhosis; end stage liver disease; sarcopenia; amino acids
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis; End Stage Liver Disease; Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXA1665 53.8 g per day (Experimental): AXA1665 administered orally TID
  Interventions: Drug: AXA1665
- Matching placebo (Placebo Comparator): Placebo administered orally TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXA1665 — AXA1665 administered TID with food
  Arms: AXA1665 53.8 g per day
Drug: Placebo — Matching placebo administered TID with food
  Arms: Matching placebo

SUMMARY:
This is a global study to compare the effects of AXA1665, an orally active mixture of amino acids, compared to placebo, on cognitive and physical function, as well as the safety and tolerability of AXA1665.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and provide written informed consent.
* Male and female adults aged ≥18 years.
* History of cirrhosis and at least 1 prior episode of overt hepatic encephalopathy (OHE) prior to Screening.
* A PHES of ≤ -4 during Screening.
* MELD score of ≤ 22 at Screening.
* Support of a primary caregiver who is able and willing to give written informed consent.

Exclusion Criteria:

* Hospitalization or serious medical condition.
* Presence of Child's-Pugh score ≥12, hepato-renal syndrome(s), refractory ascites, or spontaneous bacterial peritonitis (SBP).
* History of a surgical portosystemic or a transjugular intrahepatic portosystemic shunt (TIPS) placement.
* Expectation of a liver transplant during the study.
* Use of marijuana or tetrahydrocannabinol (THC) within 1 week prior to Screening and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in neurocognitive function by Psychometric Hepatic Encephalopathy Score (PHES) | Baseline to week 24

SECONDARY OUTCOMES:
Time to and frequency of recurrent overt hepatic encephalopathy | Baseline to week 24
Impact on physical function assessed by Liver Frailty Index (a composite measure of hand grip strength, balance and ability to stand up from a chair) | Baseline to week 24
Incidence of study product emergent adverse events (AEs) and serious adverse events (SAEs) | Baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Andres Duarte-Rojo, M.D., Principal Investigator — University of Pittsburgh
Locations (40):
- United States (21):
  - University of California, San Francisco (UCSF), San Francisco, California
  - OMEGA Research Consultants, DeBary, Florida
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - Homestead Associates in Research, Miami, Florida
  - University of Miami, Miami, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Mercy Medical Center, Baltimore, Maryland
  - New York University (NYU) School of Medicine, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Cumberland Research Associates, Fayetteville, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Optimed Research, Edinburg, Texas
  - Baylor Scott & White Research Institute, Fort Worth, Texas
  - Advanced Liver Therapies at St. Luke's Episcopal Hospital, Houston, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Bon Secours Liver Institute, Newport News, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - McGuire Research Institute, Inc., McGuire VA Medical Center, Richmond, Virginia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - LMC Diabetes & Endocrinology Ltd. - London, London, Ontario
  - The Ottawa Hospital, Ottawa
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Italy (2):
  - Azienda Ospedaliera Universitaria Federico II, Naples
  - Azienda sanitaria universitaria Friuli Centrale (ASU FC), Udine
- Poland (5):
  - KO - MED Centra Kliniczne Lublin II, Lublin
  - ID Clinic, Mysłowice
  - SONOMED Sp. z o.o., Szczecin
  - Prywatna Specjalistyczna Praktyka Lekarska Jan Gietka, Warsaw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Sp. p., Wroclaw
- Spain (6):
  - Corporacio Sanitaria Parc Tauli - Hospital de Sabadell, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
- The Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- See also: EMMPOWER Phase 2 Clinical Trial Homepage — https://emmpowertrial.com/